CLINICAL TRIAL: NCT05422898
Title: Empathic Engagement With the COVID-19 Vaccine Hesitant in Private Facebook Groups
Brief Title: Discussing COVID-19 Vaccines in Private Facebook Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCR213861
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: vaccine hesitancy; social media; health behavior
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gist (Experimental): Gist-based messages on COVID-19 vaccination and moderated group discussions in a private Facebook group
  Interventions: Behavioral: Gist messages on COVID-19 vaccination
- Information (Placebo Comparator): Link to Facebook COVID-19 Information Center
  Interventions: Behavioral: COVID-19 vaccine information

INTERVENTIONS:
Behavioral: Gist messages on COVID-19 vaccination — Participants will receive gist-based messages on COVID-19 vaccines and have their concerns addressed by a group moderator
  Arms: Gist
Behavioral: COVID-19 vaccine information — Participants will receive a link to the Facebook COVID-19 Information Center via a private Facebook Group
  Arms: Information

SUMMARY:
As the COVID-19 pandemic persists, a sizable proportion of the U.S. population remains unvaccinated and at high risk of death and serious illness from COVID-19. Vaccine hesitancy, fueled by the proliferation of vaccine misinformation on social media, is one factor contributing to lack of vaccination. Current attempts to overcome vaccine misinformation focus on correcting or debunking falsehoods. Although debunking strategies are important components to any public health campaign, communications must also address rationales for vaccine hesitancy that vary among individuals and communities, and directly address the gist of their concerns in an empathetic, non-judgmental manner. We will conduct a randomized controlled trial to test the effectiveness of empathic, relationship-building interactions relative to standard provision of information on social media to address COVID-19 vaccine hesitancy.

ELIGIBILITY:
Inclusion Criteria:

* reside in the U.S.
* unvaccinated from COVID-19
* Use Facebook regularly (at least 1/day)

Exclusion Criteria:

* age <18 years
* do not reside in the U.S.
* vaccinated from COVID-19
* do not use Facebook regularly (at least 1/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Engagement and satisfaction with the program | 4 weeks
  Engagement includes participation in the Facebook group; satisfaction=self-rated overall satisfaction with the program (7-point scale)

SECONDARY OUTCOMES:
Proportion of participants getting the COVID-19 vaccine | 4 weeks
  self-reported vaccination status
Change in COVID-19 vaccination intention | 4 weeks
  Self-reported intention to get the COVID-19 vaccine (7-point scale)
Change in intention to encourage others to get the COVID-19 vaccine | 4 weeks
  Self-reported intention to encourage others to get the COVID-19 vaccine (7-point scale)
Change in COVID-19 vaccine confidence | 4 weeks
  Self-reported confidence in the COVID-19 vaccine (5-point scale)
Change in general vaccine confidence | 4 weeks
  Self-reported confidence in vaccines (7-point scale)
Change in vaccine hesitancy | 4 weeks
  Self-reported vaccine hesitancy (7-point scale

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No